CLINICAL TRIAL: NCT07290972
Title: Compliance to Cervical Cancer Chemoradiation Guidelines: A Implementation Audit and Resource Assessment Initiative of National Cancer Grid of India
Brief Title: Compliance to Cervical Cancer Chemoradiation Guidelines: A Multicentric Implementation Audit and Resource Assessment Initiative of National Cancer Grid of India
Acronym: NCG-Compliance
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); MNJ Institute of Oncology and Regional Cancer Center (Other Government); Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor Dr Supriya Sastri, Tata Memorial Centre
Other Study IDs: TMC IEC III 900537
Record Dates: First submitted 2025-08-21; First posted 2025-12-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer Screening; Gynecologic Cancers; Treatment Compliance; Chemoradiotherapy
Keywords: Cervical cancer; Cancer; Recurrence; Treatment; Compliance; Chemoradiotherapy
MeSH Terms: conditions — Patient Compliance; Uterine Cervical Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with Cervical Cancer: Patients diagnosed with histologically proven cervical cancer wherein either radical, adjuvant or palliative radiation with or without concurrent or systemic chemotherapy planned.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Compliance to Cervical Cancer Chemoradiation treatment guidelines

SUMMARY:
This is a combination of retrospective and prospective observational study that will be performed across NCG and other participating centers to report compliance to chemoradiation for cervical cancer. This audit will include patients treated with standard of care treatment, in this case definitive or adjuvant radiation+/- concurrent chemotherapy will be included. Patients recruited in various institutions in prospective clinical trials will not be included. The participating centersthat agree to contribute data will include all registered cases over a 6-month period that have been diagnosed with cervical cancer wherein treatment is planned with radical dose radiation and/or concurrent chemotherapy. Centers that do not have retrospective data of the patients will contribute data of patients registered prospectively over 6 months. Furthermore, any cases referred to the institution for brachytherapy alone will also be included.

As a first step member institutions that participated in guideline development process or provide an agreement to guidelines adherence will be audited. The project will be submitted in institutional ethics committees with memorandum of understanding for anonymized data sharing.

Each of the co-investigators listed from contributing centers will be directly responsible for collecting data contribution and accuracy of data submitted.

Those centres which cannot or do not want to participate will be requested to provide data on only compliance outcomes to treatment for at least of 5 consecutively patients diagnosed with cervical cancer wherein treatment is planned with radical dose radiation and /or concurrent chemotherapy over a period of 6 months.

DETAILED DESCRIPTION:
Investigator intend to use electronic case record form (e-CRF) created using on line portal (google e-forms) wherein details of patients treated within the 6 month period will be captured. Google e-CRF will be available to all participating centres free of charge and has ease of access for filling details on both computer, tablets or mobile phone platforms. The e-form is user friendly and provides automated excel output and basic trends of responses and is ideal to be used across busy departments and low resource settings.

To maintain data security, no patient identifying information will be collected. Each institution will be provided an institution id and name identifiers will not be used. Similarly a code will be generated for each of the patient and details of that code will remain with the parent institution.

ELIGIBILITY:
The participating centers that agree to contribute data will include all registered cases over a 6 month period that have been diagnosed with histologically proven cervical cancer wherein either radical, adjuvant or palliative radiation with or without concurrent or systemic chemotherapy is planned.

Furthermore any cases referred to the institution for brachytherapy alone will also be included.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participating centers that agree to contribute data will include all registered cases over a 6 month period that have been diagnosed with histologically proven cervical cancer wherein either radical, adjuvant or palliative radiation with or without concurrent or systemic chemotherapy is planned.
  Furthermore any cases referred to the institution for brachytherapy alone will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 618 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
report on institutional compliance to National Cancer Grid cervical cancer guidelines for chemo-radiation. | 3 Months
  To report praportion of patients with No deviation, Major & Minor Deviation and unacceptable deviation for chemoradiation guidlines.

SECONDARY OUTCOMES:
To report on factors impacting compliance to standard guidelines | 3years
To report adequacy of infrastructural and manpower requirements for optimal treatment of cervical cancer in NCG centres and corresponding state of origin | 3 years
To compute relative risk of suboptimal treatment for cervical cancer in reference to infrastructural and manpower deficits | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Supriya Chopra, MD, Principal Investigator — ACTREC, Tata Memorial Centre, Navi Mumbai India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dr. V. K. Srivastava, Dr Tanvir Kaur, Dr. S Shrisvastava () CONSENSUS DOCUMENT FOR THE MANAGEMENT OF CANCER CERVIX, Available at: https://www.icmr.nic.in > sites > default > files > reports > Cervix Cance (Accessed: 12th December 2019).
- [Background] IAEA staffing estimator. http://nucleus.iaea.org/HHW/RadiationOncology/making the case for radiotherapy in your country/role of radiotherapy in cancer care/radiotherapy is a cost effective system which needs balance/index.html.
- [Background] IPEM recommendations for the provision of physics services to radiotherapy. http://ipem.ac.uk/portals/0/documents/recommendations.
- [Background] Budiharto T, Musat E, Poortmans P, Hurkmans C, Monti A, Bar-Deroma R, Bernstein Z, Tienhoven Gv, Collette L, Duclos F, Davis B, Aird E; EORTC Radiation Oncology Group. Profile of European radiotherapy departments contributing to the EORTC Radiation Oncology Group (ROG) in the 21st century. Radiother Oncol. 2008 Sep;88(3):403-10. doi: 10.1016/j.radonc.2008.05.013. Epub 2008 Jun 4. PMID 18538427
- [Background] International Atomic Energy Agency. Planning national radiotherapy services: a practical tool. IAEA human health series number 14. Vienna International Atomic Energy Agency;2010. ISBN 978-92-0-1059 10-9.
- [Background] Nandakumar A, Kishor Rath G, Chandra Kataki A, Poonamalle Bapsy P, Gupta PC, Gangadharan P, Mahajan RC, Nath Bandyopadhyay M, Kumaraswamy, Vallikad E, Visweswara RN, Selvaraj Roselind F, Sathishkumar K, Daniel Vijaykumar D, Jain A, Lakshminarayana Sudarshan K. Concurrent Chemoradiation for Cancer of the Cervix: Results of a Multi-Institutional Study From the Setting of a Developing Country (India). J Glob Oncol. 2015 Sep 23;1(1):11-22. doi: 10.1200/JGO.2015.000877. eCollection 2015 Oct. PMID 28804767
- [Background] Grover S, Gudi S, Gandhi AK, Puri PM, Olson AC, Rodin D, Balogun O, Dhillon PK, Sharma DN, Rath GK, Shrivastava SK, Viswanathan AN, Mahantshetty U. Radiation Oncology in India: Challenges and Opportunities. Semin Radiat Oncol. 2017 Apr;27(2):158-163. doi: 10.1016/j.semradonc.2016.11.007. Epub 2016 Nov 14. PMID 28325242
- [Background] Banerjee S, Mahantshetty U, Shrivastava S. Brachytherapy in India - a long road ahead. J Contemp Brachytherapy. 2014 Oct;6(3):331-5. doi: 10.5114/jcb.2014.45761. Epub 2014 Oct 6. PMID 25337139
- [Background] Gandhi AK, Sharma DN, Julka PK, Rath GK. Attitude and practice of brachytherapy in India: a study based on the survey amongst attendees of Annual Meeting of Indian Brachytherapy Society. J Contemp Brachytherapy. 2015 Dec;7(6):462-8. doi: 10.5114/jcb.2015.55666. Epub 2015 Nov 17. PMID 26816503
- [Background] Mittal P, Chopra S, Pant S, Mahantshetty U, Engineer R, Ghosh J, Gupta S, Ghadi Y, Menachery S, Swamidas J, Gurram L, Shrivastava SK. Standard Chemoradiation and Conventional Brachytherapy for Locally Advanced Cervical Cancer: Is It Still Applicable in the Era of Magnetic Resonance-Based Brachytherapy? J Glob Oncol. 2018 Jul;4:1-9. doi: 10.1200/JGO.18.00028. PMID 30085892
- [Background] Mahantshetty U, Krishnatry R, Hande V, Jamema S, Ghadi Y, Engineer R, Chopra S, Gurram L, Deshpande D, Shrviastava S. Magnetic Resonance Image Guided Adaptive Brachytherapy in Locally Advanced Cervical Cancer: An Experience From a Tertiary Cancer Center in a Low and Middle Income Countries Setting. Int J Radiat Oncol Biol Phys. 2017 Nov 1;99(3):608-617. doi: 10.1016/j.ijrobp.2017.06.010. Epub 2017 Jun 20. PMID 29280456
- [Background] Prescribing, Recording, and Reporting Brachytherapy for Cancer of the Cervix. J ICRU. 2013 Apr;13(1-2):NP. doi: 10.1093/jicru/ndw027. No abstract available. PMID 27335496
- [Background] Sturdza A, Potter R, Fokdal LU, Haie-Meder C, Tan LT, Mazeron R, Petric P, Segedin B, Jurgenliemk-Schulz IM, Nomden C, Gillham C, McArdle O, Van Limbergen E, Janssen H, Hoskin P, Lowe G, Tharavichitkul E, Villafranca E, Mahantshetty U, Georg P, Kirchheiner K, Kirisits C, Tanderup K, Lindegaard JC. Image guided brachytherapy in locally advanced cervical cancer: Improved pelvic control and survival in RetroEMBRACE, a multicenter cohort study. Radiother Oncol. 2016 Sep;120(3):428-433. doi: 10.1016/j.radonc.2016.03.011. Epub 2016 Apr 29. PMID 27134181
- [Background] Potter R, Tanderup K, Kirisits C, de Leeuw A, Kirchheiner K, Nout R, Tan LT, Haie-Meder C, Mahantshetty U, Segedin B, Hoskin P, Bruheim K, Rai B, Huang F, Van Limbergen E, Schmid M, Nesvacil N, Sturdza A, Fokdal L, Jensen NBK, Georg D, Assenholt M, Seppenwoolde Y, Nomden C, Fortin I, Chopra S, van der Heide U, Rumpold T, Lindegaard JC, Jurgenliemk-Schulz I; EMBRACE Collaborative Group. The EMBRACE II study: The outcome and prospect of two decades of evolution within the GEC-ESTRO GYN working group and the EMBRACE studies. Clin Transl Radiat Oncol. 2018 Jan 11;9:48-60. doi: 10.1016/j.ctro.2018.01.001. eCollection 2018 Feb. PMID 29594251
- [Background] Gupta S, Maheshwari A, Parab P, Mahantshetty U, Hawaldar R, Sastri Chopra S, Kerkar R, Engineer R, Tongaonkar H, Ghosh J, Gulia S, Kumar N, Shylasree TS, Gawade R, Kembhavi Y, Gaikar M, Menon S, Thakur M, Shrivastava S, Badwe R. Neoadjuvant Chemotherapy Followed by Radical Surgery Versus Concomitant Chemotherapy and Radiotherapy in Patients With Stage IB2, IIA, or IIB Squamous Cervical Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Jun 1;36(16):1548-1555. doi: 10.1200/JCO.2017.75.9985. Epub 2018 Feb 12. PMID 29432076
- [Background] Chopra SJ, Mathew A, Maheshwari A, Bhatla N, Singh S, Rai B, Surappa ST, Ghosh J, Sharma D, Bhaumik J, Biswas M, Deodhar K, Popat P, Giri S, Mahantshetty U, Tongaonkar H, Billimaga R, Engineer R, Grover S, Pedicayil A, Bajpai J, Rekhi B, Alihari A, Babu G, Thangrajan R, Menon S, Shah S, Palled S, Kulkarni Y, Gulia S, Naidu L, Thakur M, Rangrajan V, Kerkar R, Gupta S, Shrivastava SK. National Cancer Grid of India Consensus Guidelines on the Management of Cervical Cancer. J Glob Oncol. 2018 Jul;4:1-15. doi: 10.1200/JGO.17.00152. PMID 30085891